CLINICAL TRIAL: NCT03586466
Title: Pilot for Improved Office Based Treatment of Opioid-Dependence
Brief Title: Improving Office Based Treatment of Opioid Use Disorder With Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedicaSafe, Inc. (Industry)
Collaborators: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00023570
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Opioid-use Disorder
Keywords: opioid abuse; opioid dependence; medication assisted treatment; opioids; buprenorphine; buprenorphine/naloxone; MedicaSafe
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Micro-Electrical-Mechanical Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- BupreCare (Experimental): The BupreCare system is an integrated medication management and patient monitoring system, consisting of a smart medication-tracking dispenser and online platform. The dispensing component is a portable smart dispenser and secure pill cartridges that is programmed with an individualized treatment plan for each patient. This arm will be assigned a MedicaSafe device that will have their buprenorphine/naloxone securely stored. Treatment reports of their dispensation history will be collated and available to the treatment team.
  Interventions: Device: BupreCare; Drug: Buprenorphine/naloxone
- Treatment as Usual (Active Comparator): This arm represents an active comparator for the experimental group. Subjects in this group will undergo TAU, with no changes to the way that they receive their medication. They will have pill counts bi-weekly to examine adherence.
  Interventions: Drug: Buprenorphine/naloxone
- Treatment as Usual with MEMS (Active Comparator): This arm represents a second active comparator for the experimental group. Subjects in this group will receive their medication in a MEMS pill bottle, but otherwise will undergo TAU.
  Interventions: Drug: Buprenorphine/naloxone; Other: MEMS

INTERVENTIONS:
Device: BupreCare — Subjects will receive their medication in a MedicaSafe device. Medication will be dispensed in accordance with the programmed treatment plan for each subject. Subjects will complete a "Check-In" remotely each week with their device.
  Other Names: MedicaSafe device
  Arms: BupreCare
Drug: Buprenorphine/naloxone — Subjects will be given buprenorphine/naloxone as a component of Medication Assisted Treatment (MAT).
Other: MEMS — Subjects will receive their medication in a MEMS pill bottle.
  Arms: Treatment as Usual with MEMS

SUMMARY:
The goal of this study is to evaluate whether using a novel drug-device combination to deliver buprenorphine/naloxone (B/N) to patients in office-based treatment for Opioid Use Disorder (OUD) is an effective way to improve compliance and treatment outcomes. The system introduces psychological and behavioral supports in addition to securing the medication between doses.

DETAILED DESCRIPTION:
The misuse and abuse of opioids is a serious public health problem. SAMHSA estimates that more than 12 million Americans misuse prescription opioids for nonmedical purposes annually. The costs of this problem are substantial, both to individuals and society: total costs of prescription opioid misuse, abuse, and overdose to the US is estimated at $78.5 billion annually. Additionally, the prevalence of opioid abuse and associated costs are on the rise. In spite of this, the availability and acceptance of treatment with medications has not kept pace with the spread of the epidemic.

Prescription of buprenorphine/naloxone (B/N) is intended to address a behavioral health issue (misuse of opioids) as a component of Medication Assisted Treatment (MAT) for those who are pharmacologically dependent on opioids. In chronic illness, patient compliance and adherence with a prescribed regimen has been shown to correlate with treatment success, and conversely poor patient compliance, commonly documented, correlates with poor outcomes. Studies have demonstrated that with B/N specifically, compliance is predictive of both relapse and treatment retention. Relapse events are costly in terms of total healthcare expenditures (around $15,000 per patient), and personally - upwards of 800,000 years of potential life lost before the age of 65 in the US alone.

This study seeks to examine the effectiveness of MedicaSafe's BupreCare system in the delivery of MAT to those with OUD. The BupreCare system is a connected, locking, oral medication dispenser and secure pill cartridges coupled with an online platform. The system is programmed with a treatment plan to allow for the dispensation of medications in the right dose at the right time. Dispensation is recorded and collated in treatment reports to track patient adherence to their regimen. The project intends to ameliorate issues associated with MAT by curbing the negative effects of medication nonadherence and diversion, while simultaneously increasing provider awareness of patient behaviors and needs.

Patients aged 18-65 (inclusive) will be enrolled at Friends Research Institute in a field trial. Patients will be maintained on a stable dose of B/N, and randomized into one of three arms (BupreCare, TAU, or TAU with MEMS tracking). Subjects will have bi-weekly study visits over the course of 12 weeks. Assessments will be collected at baseline, and then every 2 weeks following study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65 years old
* Be able to provide informed consent
* Be English-speaking
* Have consistent phone and/or internet access
* Deemed by physician as medically, psychiatrically, and otherwise appropriate for buprenorphine therapy
* Maintained on a stable B/N dose

Exclusion Criteria:

* Be younger than 18 or older than 65 years of age
* Chronic pain
* Be non-English speaking
* Be unable to complete informed consent
* Be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Compliance | Compliance checks will be done every 14 days. Total compliance for each subject will be looked at across the 12-week period of participation.
  Determined by the number of days medication was taken appropriately compared to total days study medication should have been taken. For BupreCare, this will be done using the treatment reports from the device. For MEMS, this will be done with the data from the MEMS device. For TAU, this will be done with pill counts. Pill counts and dispensation reports will be supplemented by the Timeline Follow-back Assessment.

SECONDARY OUTCOMES:
Urine Drug Screens | Bi-weekly, across the 12-week participation period.
  Urine Drug Tests will be given at each in-person study visit to test for opiates and other illicit substances. The proportion of negative urine samples (for opiates) will serve as a secondary endpoint.
Relapse | Examined bi-weekly across the 12-week participation period.
  This will be determined by opiate-positive Urine Drug Screens.

OTHER OUTCOMES:
Compliance - Week 4 | Week 4 of the 12-week participation period.
  Determined by the number of days medication was taken appropriately compared to total days study medication should have been taken. For BupreCare, this will be done using the treatment reports from the device. For MEMS, this will be done with the data from the MEMS device. For TAU, this will be done with pill counts. Pill counts and dispensation reports will be supplemented by the Timeline Follow-back Assessment.
Compliance - Week 8 | Week 8 of the 12-week participation period.
  Determined by the number of days medication was taken appropriately compared to total days study medication should have been taken. For BupreCare, this will be done using the treatment reports from the device. For MEMS, this will be done with the data from the MEMS device. For TAU, this will be done with pill counts. Pill counts and dispensation reports will be supplemented by the Timeline Follow-back Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Mattai, MD, Principal Investigator — MedicaSafe, Inc.
Locations (2):
- United States (2):
  - Artemis Institute for Clinical Research, San Diego, California
  - Friends Research Institute, Baltimore, Maryland